CLINICAL TRIAL: NCT00584740
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Proof-of-concept Study to Assess the Efficacy, Safety and Tolerability of Two Single iv Infusions of AIN457 10 mg/kg (Anti IL-17 Monoclonal Antibody) in Patients With Moderate to Severe Active Crohn's Disease
Brief Title: Efficacy, Safety and Tolerability of AIN457 in Moderate to Severe Active Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely after futility criterion was met at planned interim analysis of 41 patients.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2202
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, moderate, severe, active, AIN457
MeSH Terms: conditions — Crohn Disease; Lymphoma, Follicular; Motor Activity | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIN457 (Experimental): AIN457 10 mg/kg was given as an intravenous infusion at day 1 and day 22.
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator): Matching placebo to AIN457 was given as an infusion at day 1 and day 22.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457 — 10 mg/kg
  Arms: AIN457
Drug: Placebo — Matching placebo to AIN457
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of AIN457 in patients with moderate to severe active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; 18-75 years old
* Diagnosis of Crohn's disease for at least 3 months prior to screening
* Confirmation of Crohn's disease by endoscopic or imaging examination
* Moderately active Crohn's disease at baseline, defined as:
* CDAI ≥220 and ≤450
* Active disease despite prior treatment with corticosteroids for at least 2 weeks, or immunosuppressants for at least 3 months. Treatment with azathioprine, 6-MP or MTX is allowed but must have been on a stable dose for at least 10 weeks, corticosteroids are allowed but must have been on a stable doses of prednisolone not exceeding 40 mg for two weeks prior to baseline. Immunosuppressants other than those listed above, such as cyclosporine, tacrolimus and mycophenolate, are not allowed and must be stopped (wash-out periods defined in the protocol);

Exclusion Criteria:

* Body Mass Index >34
* Positive PPD tuberculin skin test or QuantiFeron test
* Any subject with evidence of active pulmonary disease or evidence of latent tuberculosis or fungal infection at screening or within past 3 months
* Symptoms associated with active bowel structuring disease and pre-stenotic dilation on radiographs
* Fistulizing disease if complicated by sepsis and/or untreated abscess
* Multiple bowel surgeries and clinically important short bowel syndrome defined as an inability to maintain caloric intake
* Use of certain medications as specified in the protocol
* Clinical improvement due to other Crohn's therapy

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (2):
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Stuttgart

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIN457 | Placebo
Started | 39 | 20
Completed | 27 | 14
Not Completed | 12 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 8 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 | Placebo | Total
Number analyzed (Participants) | 39 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (11.96) | 38.3 (14.29) | 37.6 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 24 | 11 | 35

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Achieving Remission and/or Response
Description: Remission or response was defined as CDAI < 150 points or CDAI reduction from baseline of at least 70 points.
Time Frame: 6 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 20
Percentage of participants | 26 | 65

2. Secondary Outcome: Percentage of Participants Achieving Remission
Description: Remission was defined as CDAI < 150 points.
Time Frame: 6 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 20
Percentage of participants | 10 | 15

3. Secondary Outcome: Percentage of Participants Achieving Response
Description: Response was defined as CDAI reduction of at least 70 points from baseline.
Time Frame: 6 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 10
Percentage of participants | 26 | 65

4. Secondary Outcome: Mean Change From Baseline in CDAI Score
Description: The Crohns Disease Activity Index or CDAI is a research tool used to quantify the symptoms of patients with Crohns disease. Participants were asked to record on a paper diary the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI score: arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenousum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula; fever; use of antidiarrheal; abdominal mass; hematocrit; body weight. The CDAI score is the sum of the products of each item multiplied by its weighting factor. CDAI ranges from 0 to >=600, where remission of Crohn's disease is defined as CDAI < 150, and severe disease is defined as CDAI > 450. A negative change in mean score indicates improvement.
Time Frame: baseline, 2 weeks, 4 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 20
score on a scale
  Week 2 | -15.28 (14.010) | -52.85 (13.900)
  Week 4 | -23.52 (14.010) | -58.48 (13.900)

5. Secondary Outcome: Area Under CDAI Curve
Description: The Crohns Disease Activity Index or CDAI is a research tool used to quantify the symptoms of patients with Crohns disease. Participants were asked to record on a paper diary the frequency of stools, abdominal pain and general well-being on a daily basis. In addition to the diary data, the investigator assessed the following for the calculation of CDAI score: arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenousum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula; fever; use of antidiarrheal; abdominal mass; hematocrit; body weight. The CDAI score is the sum of the products of each item multiplied by its weighting factor. CDAI ranges from 0 to >=600, where remission of Crohn's disease is defined as CDAI < 150, and severe disease is defined as CDAI > 450. An area under the CDAI response curve analysis was performed with a starting point from week 4.
Time Frame: 10 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale*day
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 20
Units on a scale*day | 11766.26 (594.54) | 9723.45 (784.46)

6. Secondary Outcome: Percentage of Participants Maintaining Remission
Description: Remission was defined as CDAI < 150 points.
Time Frame: 10 weeks
Population: The analysis population included participants of the safety set who achieved remission.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 4 | 3
Percentage of participants | 100 | 67

7. Primary Outcome: Mean Change From Baseline in Crohns Disease Activity Index (CDAI) Score
Description: as for outcome 4
Time Frame: 6 weeks
Population: Safety Analysis Set: the safety set included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 39 | 20
score on a scale | -29.2 (14.0) | -63.1 (13.9)

ADVERSE EVENTS:
Groups:
- AIN457 Twice 10mg/kg: AIN457 10 mg/kg was given as an intravenous infusion at day 1 and day 22.
Arm/Group | AIN457 Twice 10mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 7/39 | 3/20
Other Adverse Events (participants affected / at risk) | 22/39 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Twice 10mg/kg (N=39) | Placebo (N=20)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 5 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Twice 10mg/kg (N=39) | Placebo (N=20)
Cardiac flutter (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Crohn's disease (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 5 | 1
Fatigue (General disorders) | 2 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Candidiasis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Blood pressure diastolic decreased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 3
Lethargy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.